CLINICAL TRIAL: NCT06919315
Title: Effectiveness of the Cognitive Orientation to Daily Occupational Performance (CO-OP) in a Danish Rehabilitation Context
Brief Title: Effectiveness of the Cognitive Orientation to Daily Occupational Performance (CO-OP)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Louise Møldrup Nielsen (Other)
Responsible Party: Sponsor-Investigator, Louise Møldrup Nielsen, Senior associate professor, VIA University College
Organization: VIA University College (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: CO-OP project
Record Dates: First submitted 2025-03-20; First posted 2025-04-09 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Stroke
Keywords: Stroke; Rehabilitation; CO-OP; Occupational Therapy
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: A quasi-experimental superiority trial will compare a usual practice (control) group and a CO-OP intervention group. The study will be conducted in two phases. In phase I, usual practice is delivered and in phase II, CO-OP is delivered.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental)
  Interventions: Behavioral: CO-OP intervention
- Control (Active Comparator)
  Interventions: Behavioral: Usual practice

INTERVENTIONS:
Behavioral: CO-OP intervention — CO-OP intervention: Initial phase: Goalsetting is mandatory and based on the participant's prioritized ADL performance issues identified in their baseline COPM. Education phase: Individual education in the metacognitive Goal-Plan-Do-Check strategy. Training phase: CO-OP training that involves repetitive use of the Goal-Plan-Do-Check for problem solving and skill acquisition. The therapist employs dynamic performance analysis and guided discovery to help participants understand performance issues and formulate plans for achieving their goals. Participants then execute and evaluate these plans, with a focus on developing domain-specific cognitive strategies. The therapist actively encourages generalization and transfer of skills. Homework is mandatory.
  Arms: Experimental
Behavioral: Usual practice — Usual practice: Initial phase: Goalsetting is optional and may be based on previous assessment or on a conversation with the participant. Training phase: Different approaches may be taken such as observation and practice of activities or consultation about performance issues and how participants may deal with them. The therapist may guide the participant's performance verbally, physically or trough picture materials. Homework may be included.
  Arms: Control

SUMMARY:
The goal of this clinical study is to examine the effectiveness of the Cognitive Orientation to daily Occupational Performance (CO-OP) in adults (18+) with accuired brain injury when applied in Danish rehabilitation context. The primary research question is: What is the effectiveness of the CO-OP approach on improvement of performance of daily activities (ADL) and quality of life compared to usual rehabilitation practice.

Participants in the intervention group will recieve the CO-OP intervention as part of their rehabilitation in the following phases:

Initial phase: Goalsetting is mandatory and based on the participant's prioritized ADL performance issues identified in their baseline COPM. Education phase: Individual education in the metacognitive Goal-Plan-Do-Check strategy. Training phase: CO-OP training that involves repetitive use of the Goal-Plan-Do-Check for problem solving and skill acquisition. The therapist employs dynamic performance analysis and guided discovery to help participants understand performance issues and formulate plans for achieving their goals. Participants then execute and evaluate these plans, with a focus on developing domain-specific cognitive strategies. The therapist actively encourages generalization and transfer of skills. Homework is mandatory.

Participants in the control group will recieve usual rehabilitation practice in the following phases:

Initial phase: Goalsetting is optional and may be based on previous assessment or on a conversation with the participant. Training phase: Different approaches may be taken such as observation and practice of activities or consultation about performance issues and how participants may deal with them. The therapist may guide the participant's performance verbally, physically or trough picture materials. Homework may be included.

ELIGIBILITY:
Inclusion Criteria:

* Stroke or traumatic brain injury
* Reffered from acute hospital or specialized rehabilitation units to municipal rehabilitation
* Having at least on ADL performance issue

Exclusion Criteria:

* Dementia, Psychotic diagnoses, commotio, Brain tumor or degenerative neurological conditions.
* Alkohol or drug abuse
* Not speeking or understanding Danish

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-05-02 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Canadian Occupational Performance Measure (COPM) | Baseline, up to 14 weeks, 26 weeks follow-up

SECONDARY OUTCOMES:
Assessment of Motor and Process Skills (AMPS) - ADL performance quality | Baseline, up to 14 weeks, 26 weeks follow-up
  Participants ADL performance quality will be measured with the Occupational Therapy assesment instrument, AMPS. Both process and motor skills in ADL performance will be measured and reported separately
EuroQol-5 Domain (EQ-5D-5L) | Baseline, up to 14 weeks, 26 weeks follow-up
World Health Organization Disability Assessment Schedule 2.0 (WHODAS 2.0) | Baseline, up to 14 weeks, 26 weeks follow-up
World Health Organization Quality Of Life (WHOQOL-bref) | Baseline, up to 14 weeks, 26 weeks follow-up

CONTACTS AND LOCATIONS:
Locations (2):
- Denmark (2):
  - Rehabilitation center, Skive
  - Rehabilitation center, Viborg

IPD SHARING:
Plan to Share IPD: No